CLINICAL TRIAL: NCT03255798
Title: A Prospective Evaluation of Mild to Moderate Open-Angle Glaucoma Subjects Treated With Two Second Generation Micro-bypass Stents and One Suprachoroidal Stent
Brief Title: A Prospective Evaluation of Glaucoma Subjects Treated With Two Second Generation iStents and One iStent Supra
Acronym: GCF-041
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Business decision
Sponsor: Glaukos Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GCF-041
Record Dates: First submitted 2017-08-17; First posted 2017-08-21 (Actual); Last update posted 2022-09-09 (Actual); Status verified 2022-09

CONDITIONS: Glaucoma, Open-Angle
MeSH Terms: conditions — Glaucoma, Open-Angle

STUDY DESIGN:
Intervention Model Description: G2 and G3
Masking Description: IOP outcome is masked
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- G2 and G3 implantation (Other): Two iStent inject stents and one iStent Supra stent
  Interventions: Device: G2 and G3

INTERVENTIONS:
Device: G2 and G3 — Two iStent inject devices and one iStent supra device

SUMMARY:
Prospective Evaluation of Open-Angle Glaucoma Subjects treated with two second generation iStents and one iStent Supra

DETAILED DESCRIPTION:
Prospective Evaluation of Mild to Moderate Open-Angle Glaucoma Subjects treated with Two Second Generation Microbypass Stents and One Suprachoroidal Stent

ELIGIBILITY:
Inclusion Criteria:

* Phakic or pseudophakic subjects with posterior chamber IOLs Primary open-angle glaucoma or pseudoexfoliative glaucoma diagnosis Subject on two ocular hypotensive medications Medicated screening IOP greater than or equal to 18 mm Hg and less than or equal to 30 mm Hg Visual field or optic nerve defect characteristic of glaucoma Normal iridocorneal angle anatomy Absence of peripheral anterior synechiae Mean diurnal IOP at baseline between 21 and 45 mm Hg

Exclusion Criteria:

* Subjects with anterior chamber IOLs Prior SLT or stent implantation in study eye Traumatic, uveitic, or neovascular glaucoma Fellow eye BCVA worse than 20/200

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2019-06-06 (Actual); Study Completion 2019-06-06 (Actual)

PRIMARY OUTCOMES:
20% IOP reduction | Month 12
  IOP reduction observed compared to baseline IOP, measured by Goldmann tonometry in mm Hg

SECONDARY OUTCOMES:
IOP less than or equal to 18 mm Hg | Month 12
  IOP compared to baseline IOP, measured by Goldmann tonometry in mm Hg

CONTACTS AND LOCATIONS:
Overall Officials: Kerry Stephens, OD, Study Chair — Glaukos Corporation
Locations (1):
- Prof. Dr. med. Carl Erb, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No